CLINICAL TRIAL: NCT03128190
Title: A Pragmatic Multi-center Trial of Goal-directed Fluid Management Based on Pulse Pressure Variation Monitoring During High-risk Surgery
Brief Title: Multi-center Trial of Goal-directed Fluid Management Based on Pulse Pressure Variation Monitoring
Acronym: GDTPPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Assistencia Medica ao Servidor Publico Estadual, Sao Paulo (Other)
Collaborators: University of Sao Paulo (Other); Hospital Padre Albino of Catanduva Medical School (Unknown); Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, João manoel Silva Junior, Clinical researcher, MD, PhD, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: University of Sao Paulo
Record Dates: First submitted 2017-04-11; First posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Goal-directed Fluid Therapy; Hemodynamics Instability; High-risk Surgery; Pulse-pressure Variation; Postoperative Complications
Keywords: high-risk surgery; pulse-pressure variation; monitoring; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): In the control period, patients were given intravenous fluids at the discretion of the anesthesiologist based on institutional protocol using 250ml of crystalloids or 100ml of colloids based on central venous pressure (CVP) and mean arterial pressure (MAP) measurements. The aim was to keep the CVP ≥ 8mmHg and MAP ≥ 65mmHg. Fluid boluses were administered up to a total of 1000ml, if patients did not attain a MAP of >65 mmHg, a vasopressor drug was administered.
- PPV group (Experimental): intraoperative fluid management was titrated to maintain PPV< 10%. fluids boluses of colloids were given to maintain continuously measured PPV at 10% or less
  Interventions: Other: Pulse pressure variation monitoring

INTERVENTIONS:
Other: Pulse pressure variation monitoring — fluids boluses of colloids were given to maintain continuously measured PPV at 10% or less
  Other Names: PPV
  Arms: PPV group

SUMMARY:
Background: Intraoperative fluid therapy guided by mechanical ventilation-induced pulse-pressure variation (PPV) may improve outcomes after major surgery. It was tested this hypothesis in a multi-center study.

Methods: The patients were included in two periods: a first control period (control group; n=147) in which intraoperative fluids were given according to clinical judgment. After a training period, intraoperative fluid management was titrated to maintain PPV< 10% in 109 surgical patients (PPV group). It was performed 1:1 propensity score matching to ensure the groups were comparable with regard to age, weight, duration of surgery, and type of operation. The primary endpoint was postoperative hospital length of stay.

DETAILED DESCRIPTION:
This open label, multicenter, before-and-after trial study was carried out in three hospitals, Hospital das Clínicas of São Paulo University Medical School, Hospital São Paulo of São Paulo Federal University and Hospital Padre Albino.

Subsequently obtaining IRB approval (Ethical Committee N° 0616/06 HCFMUSP) and written informed consent, high-risk patients undergoing open major surgery under general anesthesia and who required ICU admission postoperatively were enrolled from June 2007 to April 2008 (control period), followed by a phase-out period (April 2008 to July 2008) and an intervention period (July 2008 to June 2010).

High-risk surgical patients were defined as those 60 years of age or older referred to postoperative ICU care due to the presence of at least one clinical comorbidity such as coronary artery disease, chronic obstructive pulmonary disease, cerebrovascular disease, poor nutritional status, a predicted intraoperative period greater than 6 hours or predicted acute massive blood loss. All of these criteria have been used in previous studies, and they were adopted for this study. Patients with severe aortic regurgitation, cardiac arrhythmias, congestive heart failure, patients undergoing renal replacement therapy, those undergoing palliative surgery were excluded from the study.

Patients were enrolled into a standard fluid resuscitation period (Control group) or a goal-directed fluid-management group based on pulse pressure variation during the intervention period (Intervention group). Following the control period, the three-month phase-out period included education and preparation of all anesthesiology staff and logistic arrangements for the evaluation of fluid responsiveness using automated PPV measurements. Finally, the intervention period was replicated in the same season of the year as the control period.

Anesthesia care and fluid management Intraoperative monitoring standards for high-risk patients in all institutions included electrocardiography, invasive arterial blood pressure catheters, pulse oximetry, temperature monitoring, and measurement of inspiratory and expiratory gas concentrations. Additional intraoperative monitoring such as central venous catheterization was indicated on an individual basis by the attending anesthesiologist. In the interventional phase, however, intraoperative fluid adjustment was strictly directed by online PPV assessment.

In the control period, patients were given intravenous fluids at the discretion of the anesthesiologist based on institutional protocol using 250ml of crystalloids or 100ml of colloids based on central venous pressure (CVP) and mean arterial pressure (MAP) measurements. The aim was to keep the CVP ≥ 8mmHg and MAP ≥ 65mmHg. Fluid boluses were administered up to a total of 1000ml, if patients did not attain a MAP of >65 mmHg, a vasopressor drug was administered. During this initial phase, the anesthesiologists were blind to the enrollment of the patient in the study. In the interventional phase of the study, fluids boluses of colloids were given to maintain continuously measured PPV at 10% or less.

In order to evaluate PPV during surgery, an arterial line was connected to a monitor (DX 2020, Dixtal, São Paulo, SP, Brasil) specifically developed to detect respiratory variations in the arterial pressure curve, allowing for the automatic calculation of beat to beat pulse pressure, as previously described. PPV was calculated using the following formula:

PPV = 100 × (PPmax - PPmin)/[(PPmax + PPmin)/2] The mean value of PPV was automatically calculated over three consecutive floating periods of eight respiratory cycles and the median value of this triple determination was displayed on the multiparameter monitor and updated after each new respiratory cycle. The shape of the arterial curve was checked visually for damping throughout the study period. The respective hemodynamic protocols in both groups were continued until the end of surgery.

In the interventional period, the mechanical ventilator settings were adjusted using the following parameters: a) a tidal volume of 8 mL.kg-1 (ideal body weight) in volume control mode; b) an inspiratory time of 33% of the respiratory cycle; c) 5 cmH2O positive end expiratory pressure and d) respiratory rate adjusted to maintain an end-tidal capnometry of 35 mmHg to enable the measurement of PPV.

During the postoperative period, critical care and ward teams not involved in the intraoperative management or in data collection managed the patients. These individuals were not informed of patient allocation groups or study period.

Data Collection and Monitoring During the study, an investigator not participating in patient care collected all study data prospectively up until hospital discharge or patient death. Age, weight, height, sex, comorbidities such as cirrhosis, chronic obstructive pulmonary disease, hypertension, peripheral vascular disease, coronary artery disease, other cardiac disease, diabetes mellitus and cerebrovascular disease were recorded preoperatively as well as standard routine biochemical blood tests were performed. Mechanical ventilation settings, PPV values at 30 minutes' intervals, the use of vasopressors and inotropes and the duration of surgery were recorded during intraoperative. Heart rate (HR), mean arterial pressure (MAP), peripheral capillary oxygen saturation (SpO2), hemoglobin concentration and esophageal temperature were registered at the beginning and at the end of the surgical procedure. When available, central venous pressure (CVP) was recorded at the end of the surgery. The total volumes of crystalloids, colloids and blood products, percentage of patients receiving red blood cell transfusion, and use of vasopressors and inotropic drugs were recorded.

After ICU admission and 24 hours later, the following parameters were collected: HR, MAP, SpO2, CVP and arterial lactate concentration. In the ICU, the total volumes of infused crystalloids, colloids and hemocomponents were recorded as well as the percentage of patients receiving red blood cell pack (RBCP) unit transfusion. Postoperative complications were assessed daily until patient discharge according to previously published criteria: 1) vasopressor need was named circulatory shock defined by the need for continuous norepinephrine infusion after adequate fluid adjustment; 2) major ICU infections (lung, abdominal, urinary tract, line-related sepsis or wound infections); 3) respiratory dysfunction, defined as recently as recent partial pressure of oxygen in arterial blood/fraction of inspired oxygen (FiO2) of <200 without prior patient history; 4) need for reoperation; 5) need for mechanical ventilation; 6) hematologic dysfunction, defined as a platelet count of < 100,000/μL or prothrombin activity of <50%; 7) bleeding events that needed transfusion of platelets or coagulation factors; 8) • renal dysfunction, defined as a urine output of <500 mL/day, a serum creatinine level of >1.9 mg/dL, or dialysis for acute renal failure; and/or; 9) hepatic dysfunction, defined as a serum bilirubin level of >1.9 mg/dL. Postoperative length of stay and mortality were also recorded.

Upon completion of data collection from each patient, an independent Data Safety and Monitoring Board (DSMB) member conducted data quality monitoring by comparing the collected study information to the information contained in institutional medical records.

Data analysis The primary outcome of this study was postoperative length of stay. The secondary outcomes included the volume of infused fluids, RBCP transfusion, incidence of organ dysfunction, the incidence of postoperative complications and a composite outcome encompassing postoperative complications and hospital mortality rate. By using the minimal clinically significant difference between groups, eighty-one patients were required in each group to find a reduction of 2 days (from 14±5 days in the Control Group to 12±4 days in the Intervention Group), with a Type-I error of 0.05 (one-sided) and a power of 0.8.

ELIGIBILITY:
Inclusion Criteria:

* high-risk patients undergoing open major surgery under general anesthesia and who required ICU admission postoperatively

Exclusion Criteria:

* Patients with severe aortic regurgitation, cardiac arrhythmias, congestive heart failure, patients undergoing renal replacement therapy, those undergoing palliative surgery were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2007-06-01 (Actual); Primary Completion 2010-06-01 (Actual); Study Completion 2010-06-30 (Actual)

PRIMARY OUTCOMES:
postoperative length of stay | up to 90 days
  Length of hospital stay postoperatively

SECONDARY OUTCOMES:
Fluids administered postoperatively | 1 day postoperatively
  total volume of infused fluids at 24 h after ICU admission
Number of patients transfused postoperatively | 1 day postoperatively
  RBCP transfusion At 24 h after ICU admission
organ dysfunction postoperatively | up to 30 days
  incidence of organ dysfunction postoperatively (vasopressor required, mechanical ventilator required, Thrombocytopenia, Worsening liver function)
Number of patients with postoperative complications | up to 30 days
  incidence of postoperative complications (infection, reoperation, bleeding events)
hospital mortality rate | up to 30 days
  hospital mortality rate of patients

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pearse RM, Harrison DA, James P, Watson D, Hinds C, Rhodes A, Grounds RM, Bennett ED. Identification and characterisation of the high-risk surgical population in the United Kingdom. Crit Care. 2006;10(3):R81. doi: 10.1186/cc4928. Epub 2006 Jun 2. PMID 16749940
- [Result] Lobo SM, Rezende E, Knibel MF, Silva NB, Paramo JA, Nacul FE, Mendes CL, Assuncao M, Costa RC, Grion CC, Pinto SF, Mello PM, Maia MO, Duarte PA, Gutierrez F, Silva JM Jr, Lopes MR, Cordeiro JA, Mellot C. Early determinants of death due to multiple organ failure after noncardiac surgery in high-risk patients. Anesth Analg. 2011 Apr;112(4):877-83. doi: 10.1213/ANE.0b013e3181e2bf8e. Epub 2010 Jun 8. PMID 20530615
- [Result] Jhanji S, Thomas B, Ely A, Watson D, Hinds CJ, Pearse RM. Mortality and utilisation of critical care resources amongst high-risk surgical patients in a large NHS trust. Anaesthesia. 2008 Jul;63(7):695-700. doi: 10.1111/j.1365-2044.2008.05560.x. Epub 2008 May 16. PMID 18489613
- [Result] Lobo SM, Salgado PF, Castillo VG, Borim AA, Polachini CA, Palchetti JC, Brienzi SL, de Oliveira GG. Effects of maximizing oxygen delivery on morbidity and mortality in high-risk surgical patients. Crit Care Med. 2000 Oct;28(10):3396-404. doi: 10.1097/00003246-200010000-00003. PMID 11057792
- [Result] Sinclair S, James S, Singer M. Intraoperative intravascular volume optimisation and length of hospital stay after repair of proximal femoral fracture: randomised controlled trial. BMJ. 1997 Oct 11;315(7113):909-12. doi: 10.1136/bmj.315.7113.909. PMID 9361539
- [Result] Silva JM Jr, de Oliveira AM, Nogueira FA, Vianna PM, Pereira Filho MC, Dias LF, Maia VP, Neucamp Cde S, Amendola CP, Carmona MJ, Malbouisson LM. The effect of excess fluid balance on the mortality rate of surgical patients: a multicenter prospective study. Crit Care. 2013 Dec 10;17(6):R288. doi: 10.1186/cc13151. PMID 24326085
- [Result] Lopes MR, Oliveira MA, Pereira VO, Lemos IP, Auler JO Jr, Michard F. Goal-directed fluid management based on pulse pressure variation monitoring during high-risk surgery: a pilot randomized controlled trial. Crit Care. 2007;11(5):R100. doi: 10.1186/cc6117. PMID 17822565
- [Result] Auler JO Jr, Galas F, Hajjar L, Santos L, Carvalho T, Michard F. Online monitoring of pulse pressure variation to guide fluid therapy after cardiac surgery. Anesth Analg. 2008 Apr;106(4):1201-6, table of contents. doi: 10.1213/01.ane.0000287664.03547.c6. PMID 18349193
- [Result] Doherty M, Buggy DJ. Intraoperative fluids: how much is too much? Br J Anaesth. 2012 Jul;109(1):69-79. doi: 10.1093/bja/aes171. Epub 2012 Jun 1. PMID 22661747
- [Result] Suzuki S, Woinarski NC, Lipcsey M, Candal CL, Schneider AG, Glassford NJ, Eastwood GM, Bellomo R. Pulse pressure variation-guided fluid therapy after cardiac surgery: a pilot before-and-after trial. J Crit Care. 2014 Dec;29(6):992-6. doi: 10.1016/j.jcrc.2014.07.032. Epub 2014 Aug 7. PMID 25220528
- [Derived] Malbouisson LMS, Silva JM Jr, Carmona MJC, Lopes MR, Assuncao MS, Valiatti JLDS, Simoes CM, Auler JOC Jr. A pragmatic multi-center trial of goal-directed fluid management based on pulse pressure variation monitoring during high-risk surgery. BMC Anesthesiol. 2017 May 30;17(1):70. doi: 10.1186/s12871-017-0356-9. PMID 28558654
- Available data/document: Individual Participant Data Set — http://lattes.cnpq.br/0310250742582348
- Available data/document: Individual Participant Data Set — http://lattes.cnpq.br/1823080587913061